CLINICAL TRIAL: NCT04252690
Title: Physiological Study to Assess Mechanism of Action of MOBIDERM® in Lower-limb Lymphedema Patients
Acronym: ACTIODERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Collaborators: University Hospital, Tours (Other); Delta Consultants (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC18; ANSM (Other: 2019-A02043-54)
Record Dates: First submitted 2020-01-17; First posted 2020-02-05 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Lymphedema of Leg; Lymphedema Congenital; Lymphedema Primary; Lymphedema, Secondary
Keywords: lymphedema,; auto-adjustable MOBIDERM® Autofit stocking; lymphoscintigraphy; mechanism of action
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: non-randomized, open-labelled, monocentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobiderm (Experimental): MOBIDERM® autofit : auto-adjustable compression stocking
  Interventions: Device: MOBIDERM® autofit : auto-adjustable compression stocking

INTERVENTIONS:
Device: MOBIDERM® autofit : auto-adjustable compression stocking — The experimental protocol will require 2 visits during usual reduction phase performed at the hospital (5 days of hospitalization).
  Visit 1 will be performed the first day of hospitalization and will consist of inclusion visit and some evaluations (lymphoscintigraphy, edema volume, cutaneous characteristics).
  Between visit 1 (D1) and visit 2 (D3), patients will wear Mobiderm Autofit continually.
  Visit 2 will be performed the third day of hospitalization and will consist of evaluations (lymphoscintigraphy, edema volume, cutaneous characteristics, satisfaction survey).

SUMMARY:
MOBIDERM® demonstrated his interest through clinical studies on the treatment of lower or upper limb lymphedema (Mestre et al 2017; Quéré et al. 2014). This CE (Conformity European)-marking device is well established both in ambulatory and hospitalisation. Nevertheless, the mechanism of action of this device had never been confirmed and no experimental clinical studies had been performed. The hypothesis is that the MOBIDERM system creates a pressure differential between the contact zone underneath the foam cubes composing the system and their surrounding area, leading to a shear effect on the subcutaneous tissues treated.

The aim of this study is thus to assess the mechanism of action of MOBIDERM on the lymphatic system by evaluating quantitative and qualitative effects of this medical device on lymphatic system, oedema volume and cutaneous parameters in 10 lymphoedema patients during their hospitalisation for reduction phase.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary lower limb lymphedema of stage 2 or 3 according to the criteria defined by International Society of Lymphology
* Affected leg that fits with one of the standard sizes of the Auto-Adjustable MOBIDERM® Autofit stocking provided
* Signed informed consent prior to any study-mandated procedure.

Exclusion Criteria:

* Pregnant or breastfeeding patient
* Childbearing age patient without contraception
* Intolerance to Mobiderm or known allergy to the components used
* Evolutive lower limb infection
* Acute lower limb inflammation
* Dermatological ailment oozing from the treated limb
* Severe medical condition that may interfere with the proper conduct of the study
* Advanced diabetic microangiopathy
* Limb arteritis stage III or IV
* Decompensated heart failure
* Involvement in another clinical study
* Patient mentally incapable of understanding the nature, objectives and possible consequences of the study and / or refusing to submit to the constraints of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline extraction rates at 3 days after wearing MOBIDERM | Day : 3
  Assess the difference of extraction rate (%) in different areas (ankle, upper and lower middle third of the leg, knee, calf) by lymphoscintigraphy performed at D1 and D3 after wearing MOBIDERM®

SECONDARY OUTCOMES:
Change of vascular lymphatic activity between D1 and D3 | Day : 3
  Assess change of vascular lymphatic activity based on qualitative data (activity YES/NO ; quality of activity : usual - semi usual - unusual) obtained during dynamic acquisition of lymphoscintigraphy from baseline to D3
Change of lymphatic vascular flow between D1 and D3 | Day : 3
  Assess change of amplitude vascular flow : important - medium- weak ; and of flow velocity : normal, slow, inexistent from baseline to D3
Change on lymphatic system between D1 and D3 : short term effect | Day : 3
  Assess change on lymphatic system from baseline to D3 (short term effect) , based on quantitative data : number of lympho node fixation ; and qualitative data: lympho node fixation intensity : important - medium - low ; tortuous appearance of the lymphatic vessels : YES/NO ; presence of collateral : YES/NO ; presence of dermal reflux : YES/NO ; presence of popliteal ganglion : YES/NO.
Change on lymphatic system between H2 and H4 : immediate effect | Hours : 2 and 4
  Assess change on lymphatic system from baseline to 2 and 4 hours : immediate effect, based on quantitative data : number of lympho node fixation ; and qualitative data: lympho node fixation intensity : important - medium - low ; tortuous appearance of the lymphatic vessels : YES/NO ; presence of collateral : YES/NO ; presence of dermal reflux : YES/NO ; presence of popliteal ganglion : YES/NO.
Lymphedema volume reduction between D1 and D3 | Days : 1 and 3
  Leg perimeters (cm) of 7 part of leg will be measured (ankle, patella, +10cm +20cm +30cm and -10cm -20cm and -30cm of patella). Based on truncated cone formula, volume (mL) of each leg will be calculated. These volumes will be compared between D1 and D3 in order to assess lymphedema volume reduction.
Skin condition evolution between D1 and D3 | Days : 1 and 3
  Skin condition will be assessed by cutaneous ultrasound scan (skin thickness (mm) , skin echogenicity (hypoechogenicity - isoechogenicity, hyperechogenicity) , oedema distribution in the dermis (superficial dermis - deep dermis - overall of dermis -hypodermis and dermis) performed on 3 areas : ankle, leg and thigh. Skin condition evolution will be assessed at D1 and D3.
Cutaneous suppleness between D1 and D3 | Days : 1 and 3
  Cutaneous suppleness evolution is assessed with a cutometer. Cutaneous suppleness is described by skin elasticity, elastic capacity and viscoelasticity. Cutometer measurements are expressed in millimetre (skin deformation, skin relaxation, skin extensibility) and will be presented as quantitative data.
Number of type of serious and non-serious Adverse Device Effects | Day : 3
  Number and type of serious and non-serious Adverse Device Effects (ADE) will be reported during the study
Satisfaction regarding MOBIDERM | Day : 3
  Satisfaction is measured by a satisfaction questionnaire wrote specifically for the study. This questionnaire is focused on positioning the product, comfort, esthetic and global satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Loïc VAILLANT, MD, Principal Investigator — University Hospital of Tours
Locations (1):
- CHRU Tours, Tours, France

REFERENCES:
- [Background] Mestre S, Calais C, Gaillard G, Nou M, Pasqualini M, Ben Amor C, Quere I. Interest of an auto-adjustable nighttime compression sleeve (MOBIDERM(R) Autofit) in maintenance phase of upper limb lymphedema: the MARILYN pilot RCT. Support Care Cancer. 2017 Aug;25(8):2455-2462. doi: 10.1007/s00520-017-3652-5. Epub 2017 Mar 9. PMID 28281052
- [Background] Quere I, Presles E, Coupe M, Vignes S, Vaillant L, Eveno D, Laporte S, Leizorovicz A; POLIT Study investigators. Prospective multicentre observational study of lymphedema therapy: POLIT study. J Mal Vasc. 2014 Jul;39(4):256-63. doi: 10.1016/j.jmv.2014.05.004. Epub 2014 Jun 12. PMID 24931830